CLINICAL TRIAL: NCT07002346
Title: Randomized Active-controlled Trial Evaluating QL1706 Plus Bevacizumab Versus Platinum-Based Chemotherapy for Advanced First-Line Ovarian Clear Cell Carcinoma
Brief Title: INVIGORATE: A Study of QL1706 and Bevacizumab in Advanced First-Line Ovarian Clear Cell Carcinoma
Acronym: INVIGORATE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Peking Union Medical College Hospital (Other); Fudan University (Other); Sun Yat-sen University Cancer Center (SUSUCC) (Unknown); Peking University Cancer Hospital & Institute (Other); Peking University People's Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The Second Affiliated Hospital, Sun Yat-sen University (Unknown); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Renmin Hospital of Wuhan University (Other); Zhejiang Provincial People's Hospital (Other); Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); Shanghai First Maternity and Infant Hospital (Other); Hubei Cancer Hospital (Other); Sir Run Run Shaw Hospital (Other); Wuhan Central Hospital (Other); Zhejiang Cancer Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Third Affiliated Hospital of Zhengzhou University (Other); Henan Provincial People's Hospital (Other); Henan Cancer Hospital (Other Government); Jiangsu Cancer Institute & Hospital (Other); The International Peace Maternity & Child Health Hospital of China welfare institute (Unknown); Women's Hospital School Of Medicine Zhejiang University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-TJ-OCCC
Record Dates: First submitted 2025-05-20; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Clear Cell Carcinoma
Keywords: Ovarian Clear Cell Carcinoma; QL1706; Bevacizumab; First-line treatment; Immunotherapy
MeSH Terms: interventions — Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm: QL1706 + Bevacizumab (Experimental): QL1706 5 mg/kg Q3W (D1)+Bevacizumab 15mg/kg Q3W (D1) (QL1706/Bevacizumab treatment for a maximum of 2 years/22 cycles)
  Interventions: Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4); Drug: Bevacizumab
- Control Arm: Paclitaxel +Carboplatin (Active Comparator): Paclitaxel 175 mg/m2 Q3W (D1)+Carboplatin (AUC=5) Q3W (D1), 6 cycles
  Interventions: Drug: carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4) — QL1706: 5 mg/kg intravenously every 3 weeks until disease progression or intolerable toxicity, with a maximum duration of 2 years.
  Arms: Experimental Arm: QL1706 + Bevacizumab
Drug: Bevacizumab — Bevacizumab : 15 mg/kg intravenously every 3 weeks until disease progression or intolerable toxicity, with a maximum duration of 22 cycles.
  Arms: Experimental Arm: QL1706 + Bevacizumab
Drug: carboplatin — Carboplatin: AUC=5, intravenously every 3 weeks until disease progression or intolerable toxicity, with a maximum duration of 6 cycles
  Arms: Control Arm: Paclitaxel +Carboplatin
Drug: Paclitaxel — Paclitaxel: 175 mg/m^2 intravenously every 3 weeks until disease progression or intolerable toxicity, with a maximum duration of 6 cycles
  Arms: Control Arm: Paclitaxel +Carboplatin

SUMMARY:
The goal of this clinical trial is to learn if QL1706 combined with bevacizumab can effectively treat adult female patients (18 to <75 years old) with newly diagnosed FIGO stage IC-IV advanced ovarian clear cell carcinoma. The main questions it aims to answer are:

1. Does QL1706 combined with bevacizumab, compared to platinum-based chemotherapy, prolong patients' progression-free survival (PFS)?
2. What is the safety profile of QL1706 combined with bevacizumab, such as what medical problems (adverse events) do participants experience?

Researchers will compare QL1706 combined with bevacizumab (experimental arm) to a standard chemotherapy regimen of paclitaxel plus carboplatin (control arm) to see if QL1706 combined with bevacizumab is more effective in the first-line treatment of advanced ovarian clear cell carcinoma.

Participants will:

1. Be randomly assigned to receive either QL1706 combined with bevacizumab (QL1706 administered every 3 weeks, bevacizumab administered every 3 weeks) or paclitaxel plus carboplatin chemotherapy (administered every 3 weeks).
2. Visit the research center regularly for drug infusions, medical examinations (such as vital signs, physical exams, laboratory tests), and tumor imaging assessments.
3. Complete quality of life questionnaires as required.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study and signed informed consent form.
* Age ≥ 18 years and < 75 years, female.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Expected survival ≥ 3 months.
* Histologically or cytologically newly diagnosed FIGO stage IC-IV ovarian clear cell carcinoma.
* Patients who have undergone primary debulking surgery or interval debulking surgery after neoadjuvant chemotherapy, regardless of whether satisfactory debulking was achieved.
* No prior treatment with immune checkpoint inhibitors.
* Adequate organ function confirmed by the following requirements:

Hematological (no use of any blood components or cell growth factors within 7 days prior to initiation of study treatment):

i. Absolute neutrophil count (ANC) ≥ 10^9/L (1,500/mm^3). ii. Platelet count ≥ 100 × 10^9/L (100,000/mm^3). iii. Hemoglobin ≥ 90 g/L.

Renal:

i. Calculated creatinine clearance (CrCl) * ≥ 50 mL/min.

* CrCl will be calculated using the Cockcroft-Gault formula: CrCl (mL/min) = ([(140 - age) * weight (kg) * F] / [SCr (mg/dL) * 72]) Where F=0.85 (for females); SCr = serum creatinine.

ii. Urine protein < 2+ or 24-hour (h) quantitative urine protein < 1.0 g.

Hepatic:

i. Total serum bilirubin (TBil) ≤ 1.5 × ULN (Upper Limit of Normal). ii. AST (Aspartate Aminotransferase) and ALT (Alanine Aminotransferase) ≤ 2.5 × ULN.

Coagulation:

i. International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN.

- For women of childbearing potential, a negative serum or urine pregnancy test within one week prior to enrollment, and effective contraceptive measures must be used after enrollment, for example: use of physical barrier contraception (condoms) or complete abstinence. Oral, injectable, or implantable hormonal contraceptives are not permitted. Or, women of non-childbearing potential, defined as: i. Naturally postmenopausal for at least 1 year. ii. Surgically sterile (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).

iii. Serum follicle-stimulating hormone, luteinizing hormone, and plasma estradiol levels within the postmenopausal range for the study center's laboratory.

* Subject is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study requirements; patient is willing to cooperate in completing quality of life questionnaires during the trial treatment and follow-up period, and agrees that these questionnaire results can be used for clinical research.

Exclusion Criteria:

* Histologically confirmed ovarian cancer of other epithelial origin or non-epithelial origin, other than ovarian clear cell carcinoma; ovarian tumors of low malignant potential (e.g., borderline tumors).
* Prior treatment with immune checkpoint inhibitors (e.g., PD-1/PD-L1 antibodies) or drugs targeting other T-cell receptors (e.g., CTLA-4, etc.), as well as immune checkpoint agonist antibodies (e.g., anti-ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), and immune cell therapy.
* Systemic use of corticosteroids or other immunosuppressive drugs (e.g., cyclophosphamide, azathioprine, methotrexate, thalidomide, TNFα inhibitors, etc.) within 2 weeks before the first dose; Note: Inhaled or topical steroids, steroids as premedication for hypersensitivity reactions (e.g., CT scan contrast agent premedication, cytotoxic chemotherapy premedication), or adrenal replacement steroids (daily ≤10 mg prednisone or equivalent) are permitted in the absence of active autoimmune disease.
* Prior (within 5 years) or concurrent malignancies, with the exception of cured local tumors (e.g., basal cell skin cancer, squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ, breast carcinoma in situ, etc.) and breast cancer with no recurrence >3 years after radical surgery.
* Patients with contraindications to bevacizumab, including but not limited to: prior gastrointestinal perforation, surgery within 28 days before medication or incompletely healed wounds, severe bleeding or recent hemoptysis, or other situations where the investigator deems bevacizumab unsuitable.
* Receipt of live vaccine within 30 days before the first dose of study treatment (persisting until 90 days after the last dose of study treatment); Note: Live vaccines include but are not limited to measles, mumps, rubella, varicella/zoster (chickenpox), yellow fever, rabies, BCG, and typhoid vaccines. Seasonal influenza virus vaccines not containing live virus, inactivated COVID-19 vaccines, etc., are permitted.
* Active autoimmune disease requiring systemic treatment (e.g., use of disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years before the first dose. Replacement therapies (e.g., thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatment; Note: Patients with cataracts, Graves' disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Systemic infection requiring systemic antibiotic treatment or other severe infections within 2 weeks before randomization, or unexplained fever >38.0°C during the screening period or before enrollment, and inability to discontinue aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs) for more than 5 days.
* Severe illness or concomitant non-tumor diseases, such as neurological disorders, psychiatric disorders, infectious diseases, or laboratory abnormalities, that may increase the risk of participating in the study or taking study drugs, and which the investigator deems would make the patient unsuitable for the study.
* Pregnant or lactating women.
* Clinically significant cardiovascular diseases, including but not limited to:

  1. Myocardial infarction or unstable angina within 6 months before the first dose.
  2. Stroke or transient ischemic attack within 6 months before the first dose.
  3. Hypertension not controlled by optimal antihypertensive therapy (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg).
  4. Poorly controlled arrhythmias. Patients who have stabilized before the first dose and have been stable for ≥14 days may be enrolled.
  5. Congestive heart failure (New York Heart Association [NYHA] functional class II-IV).
  6. Myocarditis.
* Expectation of needing any other form of anti-tumor therapy during the study period.
* Receipt of traditional Chinese medicines with anti-tumor indications or immunomodulatory drugs (including but not limited to thymosin, interferon, interleukin-2, etc.) within 2 weeks before the first dose.
* HIV-positive patients.
* Known history of anti-tuberculosis treatment within one year before the first administration of study treatment.
* Hepatitis B surface antigen (HBsAg) positive and Hepatitis B virus DNA (HBV DNA) ≥2000 IU/ml or 10<sup>4</sup> copies/ml; HCV antibody positive and HCV RNA positive.
* Pre-existing peripheral neuropathy of grade ≥2 according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
* Current or recent (within 10 days before the first dose of study drug) continuous use of full-dose oral or parenteral anticoagulants or thrombolytic agents for 10 days (Note: Prophylactic use of low-dose anticoagulants is permitted: low-dose warfarin (≤ 1mg/d), low-dose heparin (≤ 12,000 U/d), or low-dose aspirin (≤ 100mg/d) is permitted for prophylactic purposes, provided the prothrombin time International Normalized Ratio (INR) is ≤1.5).
* Hereditary bleeding tendency or coagulation dysfunction, or history of thrombosis, or imaging showing tumor invasion/infiltration of major blood vessels, or investigator or radiologist assessment of bleeding tendency.
* Known history of severe allergy to macromolecular protein preparations, or to any component of QL1706 or other investigational drugs, or severe allergic history to chemotherapeutic drugs such as carboplatin, paclitaxel, or their premedications.
* Currently participating in interventional clinical research treatment, or receiving any other investigational drug or research device treatment within 4 weeks before the first dose (patients who failed screening for other clinical trials may be included in this study).
* Patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 4 years
  PFS is defined as the time from enrollment to the first imaging disease progression or death (whichever occurs first). Assessed according to RECIST v1.1 by BICR.

SECONDARY OUTCOMES:
Investigator-assessed PFS | Up to 4 years
  The time from enrollment to the first imaging disease progression or death (whichever occurs first). Assessed according to RECIST v1.1 by investigator.
Overall Survival (OS) | Up to 4 years
  OS is defined as the time between enrollment and the patient's death due to any cause.
Progression-Free Survival 2 (PFS2) | Up to 4 years
  Defined as the time from randomization to the second disease progression or death (whichever occurs first).
Time to First Subsequent Therapy (TFST) | Up to 4 years
  Defined as the time from the randomization date to the start date of the first subsequent anti-tumor therapy.
Time to Second Subsequent Therapy (TSST) | Up to 4 years
  Defined as the time from the randomization date to the start date of the second subsequent anti-tumor therapy.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 4 years
  Safety includes the adverse event profile of all drugs included according to the Common Terminology Criteria for Adverse Events version 5.0.

OTHER OUTCOMES:
Quality of Life (QoL) | Up to 4 years
  QoL measures the impact of the study treatment on patients' overall well-being and daily functioning, as reported by the patients themselves using standardized questionnaires like FACT-O.
Exploratory Biomarker Analysis Endpoint | Up to 4 years
  This endpoint involves analyzing various biomarkers (such as PD-L1 and TMB) from tumor tissue and blood samples to explore their potential relationship with treatment response and patient outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No